CLINICAL TRIAL: NCT02903563
Title: Knowledge Attitudes Beliefs and Practices Relative to HIV Among Sex Workers in French Guiana
Acronym: CAPProstit
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Cayenne (Other)
Responsible Party: Sponsor
Other Study IDs: CAP Prostitution
Record Dates: First submitted 2016-09-06; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: HIV
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: observational

SUMMARY:
The aim was to determine the knowledge attitudes, beliefs, and practices regarding HIV in a population of sex workers in French Guiana and in the Brazilian border town of Oiapoque. A standardized questionnaire was administered face to face to sex workers. Analysis of the questionnaires led to descriptive statistics. Multiple logistic regression models were computed to determine the predictors of condom use.

ELIGIBILITY:
Inclusion Criteria:

* sex worker

Exclusion Criteria:

* not wishing to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: sex workers
Sampling Method: Non-Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2009-01; Primary Completion 2009-01 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
knowledge attitudes practices regarding HIV and sexually transmitted diseases | when the interview was conducted
  a structured questionnaire was used. it was administered face to face with usually 5 possible responses. Scores were established using similar questions exploring related areas of HIV.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Cayenne, Cayenne, French Guiana, France

IPD SHARING:
Plan to Share IPD: No